CLINICAL TRIAL: NCT04028362
Title: Neuromuscular Blockade in the Intentive Care Unit, an Observational Study.
Acronym: CURATIV
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01378-49
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Critical Care; Mechanical Ventilation; Neuromuscular Blockade
MeSH Terms: interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuromuscular blockade: Patients who will receive neuromuscular blockade during their ICU length stay will be follow until day 28 or their hospital discharge.
  Interventions: Drug: Neuromuscular Blocking Agents

INTERVENTIONS:
Drug: Neuromuscular Blocking Agents — Patient who will receive neuromuscular blockade will be follow during their ICU lenght stay.

SUMMARY:
The study Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis. (Limit: 5000 characters) Neuromuscular blocking agents (NMBAs) are drug capable of inducing a complete paralysis of the muscle. Their use is frequent in the intensive care unit (ICU). Most of the time it is used as a single infusion to facilitate endotracheal intubation, but in the ICU the use of continuous infusion is common in several pathologies: acute distress respiratory syndrome, post-cardiac arrest survivor under hypothermia to prevent shivering, abdominal compartment syndrome, severe traumatic brain injury with uncontrolled intra-cranial pressure and severe asthma among others.

A monitoring of the dose of NMBAs is recommended to guide the depth of paralysis and to guide recovery, but in the ICU, the interest of such a monitoring during continuous infusion is unclear and the level of evidence is low.

The investigators propose to conduct a prospective multicentric observational study to describe the current practice in the use of NMBAs in mechanically ventilated patients in the ICU. As a primary objective we will describe the prevalence of NMBAs use in the ICU. As a secondary objective, the investigators will investigate the impact of protocol and/or monitoring devices of NMBAs on the dose administered and clinical outcome endpoints.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are usually administered during anesthesia for endotracheal tube placement or surgical interventions. But their use is also common in the medical intensive care unit (ICU) (1, 2). Together with sedation and analgesia, they are mainly used in continuous infusion in Acute Respiratory Distress Syndrom (ARDS) (3, 4), but also in post-cardiac arrest survivor under hypothermia to prevent shivering (5), in abdominal compartment syndrome (6), in severe traumatic brain injury with uncontrolled intra-cranial pressure (7) and severe asthma among others.

A monitoring of the treatment is recommended (8) and several monitoring techniques exists: qualitative clinical monitoring is known to be inefficient, qualitative clinical monitoring using scores such as the BSAS (9) or monitoring using peripheral nerve stimulation (train-of-four (TOF) (10)) or other devices such as accelerometry or electromyography.

As opposed to their use in the operating room where the interest of the monitoring is proven, there are discrepancy between studies on whether it is useful to monitor NMBAs in the ICU. For instance, Strange et al. did not observe any advantage of the use of a protocol of NMBAs administration (11), and Baumann et al. came to the same conclusions. However, more recently (12), Hraeich et al. found that the monitoring of NMBAs dosage guided by the TOF allowed to significantly reduce the dose administered during ADRS (13).

Thus, in the ICU, although guidelines recommend to monitor NMBAs administration (8), the level of evidence regarding the interest of monitoring and the device to use for such a monitoring is low.

The investigators propose to conduct a prospective multicentric observational study to describe the current practice in the use of NMBAs in mechanically ventilated patients in the ICU. As a primary objective the investigators will describe the prevalence of NMBAs use in the ICU. As a secondary objective, the investigator will investigate the impact of protocol and/or monitoring devices of NMBAs on the dose administered and clinical outcome endpoints, such as in-ICU mortality, duration of mechanical ventilation or acquired neuromyopathy or other complications of NMBAs.

ELIGIBILITY:
* Inclusion criteria

  * Adult Patients hospitalized in an intensive care unit
  * Patient under invasive mechanical ventilation
  * Administration of at least a single dose of neuromuscular blocking agent
* Exclusion criteria :

  * Administration of a single dose of Succinylcholine or Rocuronium for a rapid-sequence intubation
  * Moribund patient whose life expectancy is less than 24 hours
  * Patient under 18 years old
  * Patient under legal guardianship.
  * Pregnant women
  * Patient already included previously in the study
  * Absence of health insurance in France
  * Neuromuscular blocking agent administered outside the ICU (i.e. in the operating room)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in ICU and under mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who receive neuromuscular blockade | ICU Length stay (usually 7 days)
  Proportion between patients who receive neuromuscular blockade and patients hospitalized in ICU and under mechanical ventilation

SECONDARY OUTCOMES:
Indications of neuromuscular blockade | ICU Length stay (usually 7 days)
  Description of indications for neuromuscular blockade
Monitoring of neuromuscular blockade | ICU Discharge (usually 7 days)
  Proportion of patients in whom neuromuscular blockade was monitored
Neuromuscular blocking agents administered dose | ICU Discharge (usually 7 days)
  Total dose and duration of NMBAs
Tolerance of neuromuscular blocking agents | ICU Discharge (usually 7 days)
  Acquired ICU weakness, pressure ulcer, ventilator associated pneumonia, other potential side effects neuromuscular blocking agents
Number of tracheostomy | ICU Discharge (usually 7 days)
  Proportion of patients who received tracheostomy during their ICU stay
Duration of ICU stay | ICU Discharge (usually 7 days)
  Duration of ICU stay
Duration of mechanical ventilation | Time from intubation to successfull extubation (usually 5 days)
  Duration of mechanical ventilation
ICU Mortality | Time of ICU discharge (usually 7 days)
  Proportion of patients dead during their ICU length stay

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CH d'Argenteuil, Argenteuil
  - CHD Les Oudairies, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CHU Kremlin-Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU Nantes, Nantes
  - CHU Nimes, Nîmes
  - CHR Orléans, Orléans
  - CHU La Pitié Salpétrière, Paris
  - CH de Pontoise, Pontoise
  - CHRU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be obtained from PI after careful evaluation of request by clinical research committee of the French Intensive Care Society

REFERENCES:
- [Background] Arroliga A, Frutos-Vivar F, Hall J, Esteban A, Apezteguia C, Soto L, Anzueto A; International Mechanical Ventilation Study Group. Use of sedatives and neuromuscular blockers in a cohort of patients receiving mechanical ventilation. Chest. 2005 Aug;128(2):496-506. doi: 10.1378/chest.128.2.496. PMID 16100131
- [Background] Arroliga AC, Thompson BT, Ancukiewicz M, Gonzales JP, Guntupalli KK, Park PK, Wiedemann HP, Anzueto A; Acute Respiratory Distress Syndrome Network. Use of sedatives, opioids, and neuromuscular blocking agents in patients with acute lung injury and acute respiratory distress syndrome. Crit Care Med. 2008 Apr;36(4):1083-8. doi: 10.1097/CCM.0B013E3181653895. PMID 18401254
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Lascarrou JB, Le Gouge A, Dimet J, Lacherade JC, Martin-Lefevre L, Fiancette M, Vinatier I, Lebert C, Bachoumas K, Yehia A, Lagarrigue MH, Colin G, Reignier J. Neuromuscular blockade during therapeutic hypothermia after cardiac arrest: observational study of neurological and infectious outcomes. Resuscitation. 2014 Sep;85(9):1257-62. doi: 10.1016/j.resuscitation.2014.05.017. Epub 2014 Jun 2. PMID 24892266
- [Derived] Hermann B, Decormeille G, Gobe T, Mangeard N, Maamar A, Sayadi S, Pernod B, Robquin N, Ponthus JP, Le Potier S, Bouju P, Balabanian A, Frouin A, Moschietto S, Jacq G, Villemont E, Hoube C, Queyreau A, Morand C, Boissier F, Lascarrou JB, Valera S, Hraiech S, Clouet L, Piton G, Noel C, Joosten A, Tabra Osorio C, Constan A, Cecchini J, Mercier G, Bruyneel A, Villamaux C, Pousset F, Heming N, Poiroux L, Llitjos JF, Barbar SD; SRLF Trial Group. Neuromuscular blockade and their monitoring in the intensive care unit: a multicenter observational prospective study. Ann Intensive Care. 2025 Oct 22;15(1):167. doi: 10.1186/s13613-025-01591-4. PMID 41123780